CLINICAL TRIAL: NCT03520621
Title: The Role of Sulfur Amino Acids in Risk of Kwashiorkor
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: World Concern (Unknown); Action Contre la Faim (Other); Rebuild Hope for Africa (Unknown); Dignitas International (Other)
Responsible Party: Sponsor
Other Study IDs: 1605004
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Kwashiorkor
Keywords: sulfur amino acid
MeSH Terms: conditions — Kwashiorkor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Prevalence Population: Prevalence of kwashiorkor (as diagnosed by bipedal pitting edema) is >2% among children 36 to 59 months old in the population, in Murambi/Malehe Health Area of eastern Democratic Republic of the Congo
  Interventions: Other: No intervention
- Low Prevalence Population: Prevalence of kwashiorkor (as diagnosed by bipedal pitting edema) is <2% among children 36 to 59 months old in the population, in Murambi/Malehe Health Area of eastern Democratic Republic of the Congo
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
This observational cross-sectional study is investigating if young children in populations with higher prevalence of kwashiorkor malnutrition have lower dietary sulfur amino acid intake than populations with lower prevalence of kwashiorkor, controlling for multiple potential confounding factors. Intake is estimated through diet recalls during interviews with a child's caregiver, analysis of urine samples and analysis of food samples for their amino acid profiles.

DETAILED DESCRIPTION:
Kwashiorkor is one of two categorizations of severe acute malnutrition, but its etiology remains unclear. Although kwashiorkor is found only where diets are low in quality protein, comparisons of total dietary protein of individual children with and without kwashiorkor has been inconclusive. This study aims to compare amino acid profiles of the diets, not just total protein.

Evidence has shown that children with kwashiorkor consistently have very low circulating levels of sulfur amino acids (cysteine and methionine). Typical staple foods in regions with endemic kwashiorkor are generally poor in sulfur amino acids and the signs characterizing kwashiorkor can plausibly be explained by a shortage of sulfur amino acids.

In eastern Democratic Republic of the Congo, certain populations have chronically higher prevalence of kwashiorkor than neighboring populations with similar livelihoods, religion, environment, language and ethnicity. This study will compare these two populations to understand what differences between them may explain the difference in prevalence.

ELIGIBILITY:
Inclusion Criteria:

* resident of the selected population
* in the appropriate age range

Exclusion Criteria:

* caregiver reports the child has an illness that has required treatment for at least 6 months

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population, both groups, live within a 3 mile by 3 mile square in rural eastern Democratic Republic of the Congo.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-08-14 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Dietary sulfur amino acid | one measure at one time point within three weeks of registration
  mg of sulfur amino acid in the diet per kg of body weight
dietary sulfur amino acid above or below WHO estimated average requirement (EAR) | one measure at one time point within three weeks of registration
  the total sulfur amino acid in the diet will be calculated from a diet recall
  this will be a bivariate measure, "1" if the SAA in the diet is above or "0" if below the WHO/FAO requirement for sulfur amino acid intake of 17mg of sulfur amino acids per kg of body weight per day

SECONDARY OUTCOMES:
calories and protein in diet per kg of body weight | one measure at one time point within three weeks of registration
  intake of calories (kcal/kg body weight),
  digestibility adjusted protein - sum of (grams of protein per food item x digestibility of food item) per kg of body weight
  quality adjusted protein = digestibility adjusted protein in the diet x proportion of requirement of the limiting amino acid
urinary sulfate | one measure at one time point within three weeks of registration
  sulfate excreted in the urine, normalized to creatinine

OTHER OUTCOMES:
urinary thiocyanate | one measure at one time point within three weeks of registration
  thiocyanate excreted in the urine (ppm)
socio-environmental factors (use of a latrine, shelter description, feeding habits, household demographics, health history) | one measure at one time point within three weeks of registration
  sanitation - does the child use a latrine, defecate in the woods/fields, defecate around the home shelter - materials used for the roof and walls, size of the home in square meters feeding habits - number of hot meals per day, number of feeding episodes per day household demographics - age and sex of all people who eat and sleep regularly at that homestead health history - illnesses in the past 30 days, previous diagnoses of malnutrition and type of malnutrition
physical measurements of the subject's body size | one measure at one time point within three weeks of registration
  height to the nearest mm, weight to the nearest 100g, middle-upper arm circumference to the nearest mm, visual signs of kwashiorkor (edema, rough or darkened skin, friable lightened hair, distended abdomen, lethargy or irritability)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Maxwell, PhD, Principal Investigator — Tufts University, Friedman School
Locations (1):
- Restore Hope for Africa, Goma, North Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided